CLINICAL TRIAL: NCT04938076
Title: Investigation of the Effects of Noninvasive Neuromodulation in Patients With Acute Ischemic Infarction
Brief Title: Efficacy of Transcranial Direct Current Stimulation in Acute Ischemic Stroke
Acronym: DAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Collaborators: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Taewon Kim, Assistant Professor, MD, PhD, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OC19DESI0124
Record Dates: First submitted 2021-06-15; First posted 2021-06-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Double blinded randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tDCS group (Experimental): tDCS stimulation
  * affected side :
    1. primary motor cortex (M1 cortex by using the C3 or C4 position of the 10-20 EEG system)
    2. 2mA anode (+) for 30 minutes total 10 times for 7 days (ex) twice a day for 5 days)
  * contralateral unaffected side
    1. primary motor cortex (M1 cortex by using the C3 or C4 position of the 10-20 EEG system)
    2. 2mA cathode (-) for 30 minutes total 10 times for 7 days (ex) twice a day for 5 days)
  Interventions: Device: Transcranial direct current stimulation
- Sham group (Sham Comparator): . Sham stimulation
  1) the current ramps up to 2mA and slowly decreased over 30 s to ensure the typical initial tingling sensation
  Interventions: Device: sham control

INTERVENTIONS:
Device: Transcranial direct current stimulation — Transcranial direct current stimulation on motor cortex
  Arms: tDCS group
Device: sham control — sham control
  Arms: Sham group

SUMMARY:
Non-invasive brain stimulation (tDCS) such as transcranial direct current stimulation (TDCS) has been reported to be effective in improving motor performance and safe in participants with cerebral infarction. However, few studies have been done in participants with acute cerebral infarction. In this study, the investigators want to see the effect of tDCS in acute cerebral infarction. the investigators perform tDCS in participants with acute ischemic stroke within 48 hours after stroke onset and the investigators measure motor weakness and function at early phase as well as at 3 months.

DETAILED DESCRIPTION:
Cerebral infarction is a major cause of death, a disease that is socially and nationally burdensome, leaving disabilities and dementia behind.

In participants with cerebral infarction, non-invasive brain stimulation (tDCS) such as transcranial direct current stimulation (TDCS) has been reported to be effective in improving motor performance and safe. However, few studies have been done in participants with acute cerebral infarction, and previous studies in participants with acute cerebral infarction have not verified the effect in mild cerebral infarction, and previous studies in acute cerebral infarction mainly stimulate lesions to anode. So in this study, the investigators want to see the effect of stimulating tDCS to both hemispheres in acute cerebral infarction against this backdrop.

Study Objective: To see if tDCS is effective in improving motor paralysis in participants with acute cerebral infarction.

Expected effectiveness: stability of tDCS has already been demonstrated in many studies. Since tDCS itself is a non-invasive treatment, if the efficacy of the tDCS prove to be effective in patients with acute cerebral infarction, it can be widely implemented without significant risk to many patients.

Intervention : In this randomized controlled trial, the investigators perform tDCS in patients with acute ischemic stroke within 48 hours after stroke onset with sham control.

Outcome : the investigators measure motor weakness and function at early phase as well as at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* ischemic stroke patients within 2 days stroke onset
* 18-85 of age
* corticospinal tract involvement stroke (primary motor cortex, corona radiata, internal capsule, midbrain crus cerebri, basis pontis, anterior medulla)

Exclusion Criteria:

* pre-stroke disability (defined as modified Rankin Scale (mRS) >=2)
* Intravenous r-tPA thrombolysis or EVT (endovascular thrombectomy)
* history of epilepsy
* advanced systemic disease or coexisting neurological/psychiatric disease
* severe contact dermatitis or skin lesions interfering with the applying the electrode of tDCS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer (FM) motor scale, short form | at admission
  The Fugl-Meyer motor scale (FM) is widely used in clinical trials to quantify motor deficits after stroke. FM short form consists 12 items ranging from 0 (worst motor deficit) to 24 (no motor deficit).
Fugl-Meyer (FM) motor scale, short form | at 7 days
  The Fugl-Meyer motor scale (FM) is widely used in clinical trials to quantify motor deficits after stroke. FM short form consists 12 items ranging from 0 (worst motor deficit) to 24 (no motor deficit).
Fugl-Meyer (FM) motor scale, short form | at 3 month
  The Fugl-Meyer motor scale (FM) is widely used in clinical trials to quantify motor deficits after stroke. FM short form consists 12 items ranging from 0 (worst motor deficit) to 24 (no motor deficit).
NIHSS (National Institutes of Health Stroke Scale) | at admission
  National Institutes of Health Stroke Scale (NIHSS) as a Neurologic. Assessment Tool in Stroke Patients ranging from 0 (no neurologic deficit) to 42 (severe neurologic deficit).
NIHSS (National Institutes of Health Stroke Scale) | at 7 days
  National Institutes of Health Stroke Scale (NIHSS) as a Neurologic. Assessment Tool in Stroke Patients ranging from 0 (no neurologic deficit) to 42 (severe neurologic deficit).
NIHSS (National Institutes of Health Stroke Scale) | at 3 month
  National Institutes of Health Stroke Scale (NIHSS) as a Neurologic. Assessment Tool in Stroke Patients ranging from 0 (no neurologic deficit) to 42 (severe neurologic deficit).

SECONDARY OUTCOMES:
modified Rankin scale | at 3 month
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It has become the most widely used clinical outcome measure for stroke clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Taewon Kim, MD, PhD, Principal Investigator — Incheon St.Mary's Hospital
Locations (1):
- The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No